CLINICAL TRIAL: NCT04777136
Title: The Effect of Home-visit Follow-up With a Multidisciplinary Geriatric Team in Old Patients With a Hip Fracture
Brief Title: Home-visits From geRiatric tEam aFter hIp fracTure
Acronym: REFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Martin Schultz, MD, PhD, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HgH_UGT_01
Record Dates: First submitted 2021-02-16; First posted 2021-03-02 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Geriatric Assessment; Hip Fractures; Frailty; Old Age; Atrophy
Keywords: Geriatric assesment; hip fracture; Home-visit; Old patients
MeSH Terms: conditions — Hip Fractures; Frailty; Atrophy | interventions — House Calls; Geriatric Assessment; Control Groups

STUDY DESIGN:
Intervention Model Description: Home visit from the geriatric team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geriatric home visit (Experimental): Home-visit where a comprehensive geriatric assessment will be performed
  Interventions: Other: Home visit and comprehensive geriatric assessment
- Standard care (Active Comparator): No follow-up.
  Interventions: Other: Control group, no designated follow up

INTERVENTIONS:
Other: Home visit and comprehensive geriatric assessment — Home-visit from the geriatric team, who will do a full geriatric assessment and targeted interventions
  Arms: Geriatric home visit
Other: Control group, no designated follow up — Only follow-up on patients own initiative with contact to the general practitioner
  Arms: Standard care

SUMMARY:
The primary objective is to examine the effect of multidisciplinary geriatric team home-visits as follow-up after a hip fracture in old patients. The hypothesis is that home-visits will reduce the number of falls, readmissions, prevent functional decline, optimize that medical treatment, and a higher degree of satisfaction and quality of life.

DETAILED DESCRIPTION:
Among older individuals, falling is a strong predictor of frailty, morbidity, and mortality and may cause a fracture. Many older patients experience recurrent falls, further functional decline, and readmission within the first three months. Hence, fall-related visits to the hospital represent a "red flag" but are also an opportunity for targeted intervention and prevention of future falls. However, many older patients are only treated for fall-related injuries and discharged without fall risk assessment or evaluation, hence there is a need for follow-up with targeted fall assessment and intervention to prevent further falls.

Thus, the present project aims to examine the effect of home-visit follow-up of older frail patients discharged from the orthopedic ward with a hip fracture. Furthermore, we will explore the effect of a cross-sectorial collaboration between hospital and municipality in the patients' homes to prevent falls, readmissions, medicine-associated adverse effects, and physical deconditioning in old frail patients.

The present study is a interventional trial. The intervention will consist of a home visit within ten weekdays of the discharge, where a comprehensive geriatric assessment (CGA) will be performed. The team performing the CGA consist of a Geriatrician and an experienced geriatric nurse. CGA is an overall assessment of the patient taking account of; the presence and severity of comorbidity, the nutritional state, cognitive and functional status, review of current medications, and social measures. The purpose is to stabilize and optimize current as well as chronic conditions, and reduce the probability of adverse events and falls, and to secure interventions or changes persist through the transition from the secondary to the primary health care system. The assessment may lead to several interventions, including; medicine review (new medicine, change in current or discontinuation), initiation of a nutritional effort or contact to a dietitian, referral to other health care services (outpatient clinics, hospitals, or general practitioner), referral to physiotherapy and/or occupational therapy or optimization of home care.

Patients randomized to the control group will receive standard care, where the subsequent need for medical service or increased home care will require contact with the general practitioner or the municipality, at the patient's initiative.

ELIGIBILITY:
Inclusion Criteria:

* Age of 70 years or older
* Hip fracture
* Ability to provide informed consent
* Residence in one of three following municipalities: Gladsaxe, Rudersdal or Lyngby-Taarbæk

Exclusion Criteria:

* No ability to provide informed consent
* Patients, who dies within 48 hours of discharge
* Terminal patients

Nursing home residents

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to contact to the general practitioner or hospital because of a fall | 90 days
  Fall-related contact for treatment or assessment

SECONDARY OUTCOMES:
Contacts to a doctor | 90 days
  Number of contacts to a doctor (either hospital or the general practitioner)
Contacts to a doctor | 30 days
  Number of contacts to a doctor (either hospital or the general practitioner)
Falls | 30 days
  number of falls
Falls | 90 days
  number of falls
Preventable readmissions | 30 days
  Number of readmission deemed preventable by two blinded assessors
Number of drugs | 30 days
  Number of inappropriate drugs (Stop/Startt criteria)
Quality of life | 90 days
  Assessment of Quality of life using questionnaire (EQ VAS 0-100)
Patient satisfaction and fear of falling | 30 days
  Assessment patient satisfaction using questionnaire (Sat-UG-1)
Patient satisfaction and fear of faling | 90 days
  Assessment patient satisfaction using questionnaire (Sat-UG-1)
All cause mortaliy | 30 days
  Mortality
All cause mortaliy | 90 days
  Mortality
Muscle strength | 90 days
  Measured using "timed-up-and-go" test
Mobility | 90 days
  Assessed using the "new mobility score" (0-10, high is good)
Mobility | 90 days
  Assessed using the "Cumulated Ambulation Score" (0-6, high is good)
Weight | 90 days
  Change in weight i kilograms from discharge "Cumulated Ambulation Score", and "new mobility score"
Independence | 90 days
  Number of patients using walking aids
Independence | 90 days
  Number of patients with a new placement at a nursing homes

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No